CLINICAL TRIAL: NCT00136604
Title: Assess Immunogenicity, Safety & Reactogenicity of a 4th Dose of GSK Biologicals' Tritanrix-HepB/Hib-MenAC at 15-24 m & of a Dose of Mencevax ACWY at 24-30 m in Subjects Primed With 3 Doses of Tritanrix-HepB/Hib-MenAC
Brief Title: Response to GSK Biologicals' Tritanrix-HepB/Hib-MenAC Vacc (4th Dose) at 15-24m & Mencevax ACWY at 24-30m
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104727 (Booster - 15-24 mths); 104730
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Whole Cell Pertussis; Haemophilus Influenzae Type b; Hepatitis B; Diphtheria; Tetanus; Diphtheria-Tetanus-Pertussis-Hepatitis B-Haemophilus Influenzae Type b-Neisseria Meningitidis Vaccin
Keywords: Prophylaxis diphtheria; Hib & meningococcal serogroup A & C disease
MeSH Terms: conditions — Haemophilus Infections; Hepatitis B; Diphtheria; Tetanus | interventions — PsACWY vaccine

STUDY DESIGN:
Who Masked: Care Provider

ARMS (5):
- ACAC GROUP (Experimental): Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine in the primary study (NCT00317161) are boosted in the current study with one dose of the same vaccines at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age.
  Interventions: Biological: Tritanrix-HepB/Hib-MenAC
- ACHibPS GROUP (Experimental): Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with MenAC-TT vaccine in the primary study (NCT00317161) are boosted in the current study with one dose of Tritanrix-HepB/Hiberix at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Mencevax ACWY; Biological: Tritanrix-HepB/Hiberix
- HibACPS GROUP (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317161) are boosted in the current study with one dose of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
  Interventions: Biological: Tritanrix-HepB/Hib-MenAC; Biological: Mencevax ACWY
- HibHibPS GROUP (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317161) are boosted in the current study with one dose of the same vaccine at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects are also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
  Interventions: Biological: Mencevax ACWY; Biological: Tritanrix-HepB/Hiberix
- CC GROUP (Experimental): Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix + Meningitec vaccine in the primary study (NCT00317161) are boosted in the current study with one dose of the same vaccine at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age.
  Interventions: Biological: Tritanrix-HepB/Hiberix; Biological: Meningitec

INTERVENTIONS:
Biological: Tritanrix-HepB/Hib-MenAC — Combined Diphtheria, Tetanus, Whole Cell Pertussis, Hepatitis B, Haemophilus influenzae Type b meningococcal AC-tetanus toxoid conjugate Vaccine
  Arms: ACAC GROUP; HibACPS GROUP
Biological: Mencevax ACWY — GSK Biologicals' Meningococcal serogroups A, C, W135 and Y polysaccharide vaccine
  Arms: ACHibPS GROUP; HibACPS GROUP; HibHibPS GROUP
Biological: Tritanrix-HepB/Hiberix — Combined Diphtheria, Tetanus, Whole Cell Pertussis, Hepatitis B Vaccine, Haemophilus influenzae type b conjugate vaccine
  Arms: ACHibPS GROUP; CC GROUP; HibHibPS GROUP
Biological: Meningitec — Wyeth's MenC CRM197 conjugated vaccine, Meningitec
  Arms: CC GROUP

SUMMARY:
The purpose of the study is to evaluate the immunogenicity, safety and reactogenicity of a booster dose of DTPw-HBV/Hib-MenAC compared to DTPw-HBV/Hib given to healthy subjects at 15 to 24 months of age primed with 3 doses of Tritanrix-HepB/Hib-MenAC in study 100480. Antibody persistence will be evaluated at 24 to 30 months. Immunogenicity, safety and reactogenicity of a dose of Mencevax ACWY given at 24 to 30 months will also be evaluated when given to subjects not boosted with a MenA conjugate and/or MenC containing vaccine.

DETAILED DESCRIPTION:
This study will be conducted in two stages. In the DTP booster phase subjects will receive a booster dose of Tritanrix-HepB/Hib-MenAC or Tritanrix-HepB/Hib (active control) at 15 to 24 months in a single-blind manner so that the subjects' parents will not know which vaccine was administered to their child (this booster phase is no longer recruiting). In the Mencevax ACWY phase at 24-30 months a dose of Mencevax ACWY will be given to subjects who were not boosted with a MenA conjugate and/or MenC containing vaccine at 15-24 months in an open manner (this booster phase is not yet recruiting). Up to four blood samples will be taken: before and one month after the administration of the DTP booster dose and of Mencevax ACWY. To comply with the immunisation calender of Thailand, at 15-24 months all subjects will receive OPV. At 16-25 months 2 doses of Japanese Encephalitis (JE) vaccine or a dose of varicella vaccine will be offered and at 25-31 months a dose of varicella or JE vaccine will be offered.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female between and including 15 and 24 months of age
* Having participated in the primary vaccination study DTPW-HBV=HIB-MENAC-TT-003 (eTrack No. 100480)

Exclusion criteria:

* Booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b (Hib) and/or meningococcal serogroups A and/or C disease not foreseen in the protocol, after the date of the study conclusion visit of the primary vaccination study DTPW-HBV=HIB-MENAC-TT-003 (eTrack No. 100480).
* History of or known exposure to diphtheria, tetanus, pertussis, hepatitis B, Hib and/or meningococcal serogroup A or C disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures including febrile seizures (at least two events) in infancy.

Ages: 427 Days to 730 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 617 (Actual)
Dates: Start 2006-01-22 (Actual); Primary Completion 2006-04-23 (Actual); Study Completion 2006-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Primary Study — http://www.clinicaltrials.gov/ct/show/NCT00317161
- Available data/document: Individual Participant Data Set: 104727 (Booster - 15-24 mths) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104727 (Booster - 15-24 mths) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104727 (Booster - 15-24 mths) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104727 (Booster - 15-24 mths) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104727 (Booster - 15-24 mths) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104727 (Booster - 15-24 mths) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- ACAC GROUP: Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine in the primary study (NCT00317161) were boosted in the current study with one dose of the same vaccines at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age.
- ACHibPS GROUP: Subjects vaccinated with 3 doses of Tritanrix-Hepb co-administrated with MenAC-TT vaccine in the primary study (NCT00317161) were boosted in the current study with one dose of Tritanrix-HepB/Hiberix at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
- HibACPS GROUP: Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317161) were boosted in the current study with one dose of Tritanrix-Hepb co-administrated with Hib-MenAC-TT vaccine at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm
- HibHibPS GROUP: Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix vaccine in the primary study (NCT00317161) were boosted in the current study with one dose of the same vaccine at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. Subjects were also administered one booster dose of Mencevax ACWY vaccine at 24 to 30 months of age by deep subcutaneous injection in the upper region of the left arm.
- CC GROUP: Subjects vaccinated with 3 doses of Tritanrix-HepB/Hiberix + Meningitec vaccine in the primary study (NCT00317161) were boosted in the current study with one dose of the same vaccine at 15 to 24 months of age, intramuscularly into the anterolateral quadrant of the left thigh or upper region of the left arm. No Mencevax ACWY vaccine at 24 to 30 months of age.
Period: Overall Study
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Started | 249 | 123 | 79 | 41 | 125
Completed | 248 | 122 | 79 | 41 | 124
Not Completed | 1 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1
Not completed — Migrated/moved from study area | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP | Total
Number analyzed (Participants) | 249 | 123 | 79 | 41 | 125 | 617
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.90 (0.52) | 17.8 (0.59) | 17.7 (0.59) | 17.7 (0.67) | 17.8 (0.55) | 17.82 (0.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 56 | 38 | 21 | 55 | 302
  Male | 117 | 67 | 41 | 20 | 70 | 315
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Information about race distribution was not available in the report; it was obtained from the primary study.
  Participants
    East - South East Asian | 249 | 123 | 79 | 41 | 125 | 617

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Meningococcal C Serum Bactericidal Assay (SBA-MenC) Antibody Titers Above the Cut-off Value
Description: Pre-defined assay cut-off value for assessed titers was greater than or equal to (≥) 1:128.
Time Frame: One month Post-Booster vaccination at 15-24 months of age
Population: The Booster According-to-Protocol (ATP) cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available.This primary analysis focused only on subjects from Tritanrix-Hepb/Hib-MenAC-TT Group versus TRITANRIX-HEPB+Mencevax + Meningitec Group.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | CC GROUP
Number analyzed (Participants) | 247 | 122
Percentage | 100 | 100
Statistical Analysis 1: Comparison: ACAC GROUP vs CC GROUP; Demonstration of non-inferiority of a fourth dose of the Tritanrix-HepB/Hib-MenAC-TT vaccine versus a fourth dose of the Tritanrix-HepB/Hiberix and Meningitec vaccine given concomitantly in terms of the percentage of subjects with an SBA-MenC titre ≥ 1:128; Test type: Non-Inferiority — Criterion for non-inferiority evaluation: The lower limit (LL) of the standardized asymptotic 95% confidence interval (CI) on the difference in the percentage of subjects with SBA-MenC titre ≥ 1:128 between the Tritanrix-Hepb/Hib-MenAC-TT Group and (minus) the TRITANRIX-HEPB+Mencevax + Meningitec control group was above -10%; Difference in percentage of subjects = 0.00, 95% CI 2-sided [-1.53 to 3.05]

2. Primary Outcome: Percentage of Subjects With SBA-MenA Antibody Titers Above the Cut-off Value
Description: Pre-defined assay cut-off value for assessed titers was greater than or equal to (≥) 1:128. Note: For the MenA antibodies with assay on SBA, additional testing were done using a serogroup A strain 3125 (L10 immunotype).
Time Frame: One Month Post-Booster vaccination at 15-24 months of age
Population: The Booster According-to-Protocol (ATP) cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available. This primary analysis focused on subjects from Tritanrix-Hepb/Hib-MenAC-TT Group only.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP
Number analyzed (Participants) | 224
Percentage
  rSBA-MenA (L11): number analyzed (Participants) | 136
  rSBA-MenA (L11) | 100
  rSBA-MenA (L10) | 100

3. Primary Outcome: Percentage of Seroprotected (SPR) Subjects With Anti-Polyribosyl Ribitol Phosphate Anti-(PRP) Antibody Concentrations Above the Cut-off Value
Description: Antibody concentrations cut-off value was ≥ 1 microgram per milliliter (µg/mL).
Time Frame: One Month Post-Booster vaccination at 15-24 months of age
Population: The Booster ATP cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available. This primary analysis focused only on subjects from Tritanrix-Hepb/Hib-MenAC-TT versus Tritanrix-Hepb/Mencevax+Tritanrix-HepB/Hiberix groups.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | ACHibPS GROUP
Number analyzed (Participants) | 247 | 122
Percentage | 100 | 100
Statistical Analysis 1: Comparison: ACAC GROUP vs ACHibPS GROUP; Demonstration of non-inferiority of the Tritanrix-HepB/Hib-MenAC-TT vaccine versus the Tritanrix-HepB/Hiberix vaccine when used as a booster vaccine in Tritanrix-HepB/Hib-MenAC-TT primed subjects in terms of the percentage of subjects with an anti-PRP concentration ≥ 1.0 µg/mL; Test type: Non-Inferiority — Criterion for non-inferiority evaluation: The lower limit (LL) of the standardized asymptotic 95% CI on the difference in seroprotection (anti-PRP concentration ≥ 1.0 µg/mL) between the Tritanrix-Hepb/Hib-MenAC-TT Group and (minus) the Tritanrix-Hepb/Mencevax+Tritanrix-HepB/Hiberix Group was above -10%; Difference in seroprotection rate = 0.00, 95% CI 2-sided [-1.53 to 3.05]

4. Secondary Outcome: Percentage of SPR Subjects With Anti-(PRP) Antibody Concentrations Above Predefined Cut-off Values
Description: Antibody concentrations cut-off values were ≥ 0.15 and ≥ 1 micrograms per milliliter (µg/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: The Booster According-to-Protocol (ATP) cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 247 | 122 | 76 | 41 | 122
Percentage
  Anti-PRP ≥ 0.15 µg/mL (Pre-Booster) | 100 | 99.2 | 100 | 100 | 99.2
  Anti-PRP ≥ 0.15 µg/mL (Post-Booster) | 100 | 100 | 100 | 100 | 100
  Anti-PRP ≥ 1 µg/mL (Pre-Booster) | 88.3 | 86.1 | 88.2 | 87.8 | 89.3
  Anti-PRP ≥ 1 µg/mL (Post-Booster) | 100 | 100 | 100 | 100 | 100

5. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as Geometric Mean Concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 247 | 122 | 76 | 41 | 122
μg/mL
  Anti-PRP (Pre-Booster) | 4.572 [3.859 to 5.416] | 4.371 [3.411 to 5.602] | 3.728 [2.872 to 4.840] | 4.498 [3.144 to 6.436] | 4.775 [3.774 to 6.041]
  Anti-PRP (Post-Booster) | 85.798 [75.274 to 97.793] | 168.232 [140.939 to 200.812] | 56.772 [44.788 to 71.962] | 129.222 [95.254 to 175.301] | 115.384 [95.550 to 139.336]

6. Secondary Outcome: Percentage of Subjects With SBA-MenC Antibody Titers Above the Cut-off Values
Description: Pre-defined assay cut-off values for assessed titers were greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: The Booster ATP cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available. This analysis focused only on subjects from groups boosted with a vaccine containing a MenC conjugate.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | HibACPS GROUP | CC GROUP
Number analyzed (Participants) | 247 | 76 | 122
Percentage
  Anti-SBA-MENC ≥ 1:8 (Pre-Booster): number analyzed (Participants) | 246 | 75 | 119
  Anti-SBA-MENC ≥ 1:8 (Pre-Booster) | 95.1 | 10.7 | 90.8
  Anti-SBA-MENC ≥ 1:8 (Post-Booster) | 100 | 100 | 100
  Anti-SBA-MENC ≥ 1:128 (Pre-Booster): number analyzed (Participants) | 246 | 75 | 119
  Anti-SBA-MENC ≥ 1:128 (Pre-Booster) | 82.1 | 8.0 | 61.3
  Anti-SBA-MENC ≥1:128 (Post-Booster) | 100 | 100 | 100

7. Secondary Outcome: Anti-SBA-MenC Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ACAC GROUP | HibACPS GROUP | CC GROUP
Number analyzed (Participants) | 247 | 76 | 122
Titers
  Anti-SBA-MenC (Pre-Booster): number analyzed (Participants) | 246 | 75 | 119
  Anti-SBA-MenC (Pre-Booster) | 295.2 [245.7 to 354.6] | 6.3 [4.6 to 8.7] | 143.8 [105.3 to 196.4]
  Anti-SBA-MenC (Post-Booster) | 4891.2 [4466.0 to 5356.9] | 1868.4 [1495.0 to 2335.0] | 8068.6 [6717.7 to 9691.3]

8. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Assay Against Meningococcal Serogroup A Using Rabbit Complement (rSBA-MenA) Antibody Titers Above the Pre-defined Cut-off Values
Description: Pre-defined assay cut-off values for assessed titers were greater than or equal to (≥) 1:8 and (≥) 1:128. Note: For the MenA antibodies with assay on SBA, additional testing were done using a serogroup A strain 3125 (L10 immunotype).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: The Booster ATP cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available. This analysis focused only on subjects from groups boosted with a vaccine containing a MenA conjugate.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | HibACPS GROUP | HibHibPS GROUP
Number analyzed (Participants) | 226 | 74 | 38
Percentage
  rSBA-MenA (L11) ≥ 1:8 Pre-Booster: number analyzed (Participants) | 226 | 70 | 34
  rSBA-MenA (L11) ≥ 1:8 Pre-Booster | 99.6 | 88.6 | 94.1
  rSBA-MenA (L11) ≥ 1:8 Post-Booster: number analyzed (Participants) | 136 | 74 | 38
  rSBA-MenA (L11) ≥ 1:8 Post-Booster | 100 | 100 | 97.4
  rSBA-MenA (L11) ≥ 1:128 Pre-Booster: number analyzed (Participants) | 226 | 70 | 34
  rSBA-MenA (L11) ≥ 1:128 Pre-Booster | 96.9 | 85.7 | 94.1
  rSBA-MenA (L11) ≥1:128 Post-Booster: number analyzed (Participants) | 136 | 74 | 38
  rSBA-MenA (L11) ≥1:128 Post-Booster | 100 | 100 | 97.4
  rSBA-MenA (L10) ≥ 1:8 Pre-Booster: number analyzed (Participants) | 224 | 59 | 33
  rSBA-MenA (L10) ≥ 1:8 Pre-Booster | 88.8 | 54.2 | 57.6
  rSBA-MenA (L10) ≥ 1:8 Post-Booster: number analyzed (Participants) | 224 | 73 | 30
  rSBA-MenA (L10) ≥ 1:8 Post-Booster | 100 | 100 | 90.0
  rSBA-MenA (L10) ≥ 1:128 Pre-Booster: number analyzed (Participants) | 224 | 59 | 33
  rSBA-MenA (L10) ≥ 1:128 Pre-Booster | 66.1 | 42.4 | 42.4
  rSBA-MenA (L10) ≥ 1:128 Post-Booster: number analyzed (Participants) | 224 | 73 | 30
  rSBA-MenA (L10) ≥ 1:128 Post-Booster | 100 | 100 | 70.0

9. Secondary Outcome: Anti-rSBA-MenA Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ACAC GROUP | HibACPS GROUP | HibHibPS GROUP
Number analyzed (Participants) | 246 | 76 | 122
Titers
  rSBA-MenA (L11), Pre-Booster: number analyzed (Participants) | 246 | 70 | 34
  rSBA-MenA (L11), Pre-Booster | 626.2 [551.6 to 711.0] | 327.2 [215.4 to 497.0] | 468.3 [290.3 to 755.4]
  rSBA-MenA (L11), Post-Booster: number analyzed (Participants) | 136 | 74 | 38
  rSBA-MenA (L11), Post-Booster | 1488.8 [1318.7 to 1680.8] | 3429.6 [2939.5 to 4001.4] | 411.5 [297.0 to 570.0]
  rSBA-MenA (L10), Pre-Booster: number analyzed (Participants) | 224 | 59 | 33
  rSBA-MenA (L10), Pre-Booster | 141.1 [115.1 to 172.9] | 37.1 [21.3 to 64.7] | 33.8 [17.1 to 67.0]
  rSBA-MenA (L10), Post-Booster: number analyzed (Participants) | 224 | 73 | 30
  rSBA-MenA (L10), Post-Booster | 1784.8 [1611.2 to 1977.1] | 1663.7 [1415.4 to 1955.6] | 172.5 [100.4 to 296.3]

10. Secondary Outcome: Percentage of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentrations Above the Predefined Cut-off Values
Description: Antibody concentrations cut-off values were ≥ 0.3 and ≥ 2 micrograms per milliliter (µg/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 6
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | HibACPS GROUP | CC GROUP
Number analyzed (Participants) | 247 | 76 | 122
Percentage
  Anti-PSC ≥ 0.3 µg/mL (Pre-Booster) | 97.2 | 3.9 | 97.5
  Anti-PSC ≥ 0.3 µg/mL (Post-Booster): number analyzed (Participants) | 246 | 76 | 122
  Anti-PSC ≥ 0.3 µg/mL (Post-Booster) | 100 | 100 | 100
  Anti-PSC ≥ 2 µg/mL (Pre-Booster) | 33.6 | 1.3 | 30.3
  Anti-PSC ≥ 2 µg/mL (Post-Booster): number analyzed (Participants) | 246 | 76 | 122
  Anti-PSC ≥ 2 µg/mL (Post-Booster) | 99.2 | 100 | 100

11. Secondary Outcome: Anti-PSC Antibody Concentrations
Description: Antibody concentrations were presented as Geometric Mean Concentrations (GMCs) and expressed in micrograms/milliliter (µg/ml).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/ml
Arm/Group | ACAC GROUP | HibACPS GROUP | CC GROUP
Number analyzed (Participants) | 247 | 76 | 122
µg/ml
  Anti-PSC (Pre-Booster) | 1.37 [1.24 to 1.53] | 0.16 [0.15 to 0.18] | 1.41 [1.23 to 1.62]
  Anti-PSC (Post-Booster): number analyzed (Participants) | 246 | 76 | 122
  Anti-PSC (Post-Booster) | 11.71 [10.82 to 12.68] | 25.96 [22.73 to 29.65] | 31.42 [27.29 to 36.17]

12. Secondary Outcome: Percentage of Subjects With Anti-polysaccharide A (Anti-PSA) Antibody Concentrations Above the Predefined Cut-off Values
Description: Antibody concentrations cut-off values were ≥ 0.3 and ≥ 2 micrograms per milliliter (µg/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 8
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | HibACPS GROUP | HibHibPS GROUP
Number analyzed (Participants) | 246 | 76 | 41
Percentage
  Anti-PSA ≥ 0.3 µg/ml (Pre-Booster) | 78.9 | 18.4 | 7.3
  Anti-PSA ≥ 0.3 µg/ml (Post-Booster): number analyzed (Participants) | 246 | 76 | 40
  Anti-PSA ≥ 0.3 µg/ml (Post-Booster) | 100 | 100 | 15.0
  Anti-PSA ≥ 2 µg/ml (Pre-Booster) | 12.6 | 2.6 | 2.4
  Anti-PSA ≥ 2 µg/ml (Post-Booster): number analyzed (Participants) | 246 | 76 | 40
  Anti-PSA ≥ 2 µg/ml (Post-Booster) | 97.6 | 100 | 0.0

13. Secondary Outcome: Anti-PSA Antibody Concentrations
Description: Antibody concentrations were presented as Geometric Mean Concentrations (GMCs) ad expressed in micrograms per milliliter ().
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: µg/ml
Arm/Group | ACAC GROUP | HibACPS GROUP | HibHibPS GROUP
Number analyzed (Participants) | 246 | 76 | 41
µg/ml
  Anti-PSA (Pre-Booster) | 0.64 [0.57 to 0.72] | 0.20 [0.17 to 0.23] | 0.17 [0.15 to 0.20]
  Anti-PSA (Post-Booster): number analyzed (Participants) | 246 | 76 | 40
  Anti-PSA (Post-Booster) | 20.31 [17.92 to 23.01] | 14.20 [11.95 to 16.88] | 0.19 [0.16 to 0.23]

14. Secondary Outcome: Percentage of Seroprotected (SPR) Subjects With Anti-diphtheria Toxoid (Anti-DT) Antibody Concentrations Above the Predefined Cut-off Values
Description: Antibody concentrations cut-off values were ≥ 0.1 international units per milliliter (IU/mL) as assessed by enzyme-linked immunosorbent assay (ELISA) or ≥ 0.016 IU/ml as assessed by Vero cell neutralization test if concentrations were < 0.1 IU/ml when assessed by ELISA.
Time Frame: One month after (POST) the Booster vaccination at 15-24 months of age
Population: The Booster ATP cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence and for whom data concerning the immunogenicity measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after the booster vaccination.
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 120 | 119 | 76 | 41 | 117
Percentage | 99.2 | 100 | 100 | 100 | 100

15. Secondary Outcome: Anti-D Antibody Concentrations
Description: Antibody concentrations were presented as Geometric Mean Concentrations (GMCs) and expressed in international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: The Booster ATP cohort for Immunogenicity included all evaluable subjects from the Booster ATP cohort for Persistence, for whom data concerning the immunogenicity measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component pre/after the booster vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 120 | 119 | 76 | 41 | 117
IU/mL
  Anti-D (Pre-Booster): number analyzed (Participants) | 119 | 119 | 76 | 41 | 117
  Anti-D (Pre-Booster) | 0.126 [0.105 to 0.150] | 0.137 [0.116 to 0.162] | 0.134 [0.108 to 0.166] | 0.124 [0.091 to 0.169] | 0.168 [0.143 to 0.198]
  Anti-D (Post-Booster) | 4.705 [3.714 to 5.962] | 5.003 [3.958 to 6.324] | 5.297 [3.968 to 7.070] | 5.777 [3.625 to 9.205] | 9.269 [7.812 to 10.997]

16. Secondary Outcome: Percentage of Seroprotected (SPR) Subjects With Anti-tetanus Toxoid (Anti-TT) Antibody Concentrations Above the Predefined Cut-off Values
Description: Antibody concentrations cut-off value was ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 15
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 120 | 119 | 76 | 41 | 117
Percentage
  Anti-TT (Pre-Booster) | 99.2 | 99.2 | 97.4 | 97.6 | 96.6
  Anti-TT (Post-Booster) | 100 | 100 | 100 | 100 | 100

17. Secondary Outcome: Anti-TT Antibody Concentrations
Description: as for outcome 15
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 120 | 119 | 76 | 41 | 117
IU/mL
  Anti-TT (Pre-Booster) | 0.709 [0.622 to 0.809] | 0.648 [0.570 to 0.737] | 0.617 [0.519 to 0.735] | 0.537 [0.427 to 0.675] | 0.566 [0.489 to 0.655]
  Anti-TT (Post-Booster) | 16.313 [15.089 to 17.636] | 18.942 [17.203 to 20.857] | 12.531 [10.902 to 14.405] | 13.125 [11.071 to 15.560] | 10.792 [9.618 to 12.108]

18. Secondary Outcome: Percentage of Seroprotected (SPR) Subjects With Anti-Bordetella Pertussis Toxoid (Anti-BPT) Antibody Concentrations Above the Predefined Cut-off Value
Description: Antibody concentrations cut-off value was ≥ 15 ELISA units per milliliter (EL.U/mL).
Time Frame: One month Post-Booster vaccination
Population: as for outcome 14
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 114 | 111 | 69 | 38 | 110
Percentage | 98.2 | 100 | 100 | 97.4 | 99.1

19. Secondary Outcome: Anti-BPT Antibody Concentrations
Description: Antibody concentrations were presented as Geometric Mean Concentrations (GMCs) and expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/ml
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 118 | 117 | 74 | 40 | 117
EL.U/ml
  Anti-BPT (Pre-Booster) | 11.7 [10.3 to 13.3] | 10.5 [9.5 to 11.7] | 10.6 [9.2 to 12.3] | 10.5 [8.8 to 12.6] | 11.1 [9.9 to 12.4]
  Anti-BPT (Post-Booster): number analyzed (Participants) | 116 | 113 | 71 | 39 | 110
  Anti-BPT (Post-Booster) | 122.1 [109.8 to 135.8] | 115.9 [105.1 to 127.9] | 129.1 [114.0 to 146.2] | 112.6 [90.0 to 140.8] | 102.5 [92.4 to 113.7]

20. Secondary Outcome: Percentage of Seroprotected (SPR) Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentrations Above the Predefined Cut-off Value
Description: Antibody concentrations cut-off value was ≥ 10 international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 15
Measure: Number; unit: Percentage
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 120 | 119 | 76 | 41 | 116
Percentage
  Anti-HBs (Pre-Booster): number analyzed (Participants) | 115 | 119 | 76 | 41 | 114
  Anti-HBs (Pre-Booster) | 82.6 | 90.8 | 94.7 | 90.2 | 81.6
  Anti-HBs (Post-Booster): number analyzed (Participants) | 120 | 119 | 76 | 40 | 116
  Anti-HBs (Post-Booster) | 95.8 | 97.5 | 98.7 | 100 | 96.6

21. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as Geometric Mean Concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: Prior to (PRE) and one month after (POST) the Booster vaccination at 15-24 months of age
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 120 | 119 | 76 | 41 | 116
mIU/ml
  Anti-HBs (Pre-Booster): number analyzed (Participants) | 115 | 119 | 76 | 41 | 114
  Anti-HBs (Pre-Booster) | 54.8 [41.3 to 72.8] | 91.2 [71.8 to 115.7] | 95.0 [71.1 to 126.8] | 84.4 [55.3 to 129.0] | 65.6 [48.9 to 88.2]
  Anti-HBs (Post-Booster): number analyzed (Participants) | 120 | 119 | 76 | 40 | 116
  Anti-HBs (Post-Booster) | 3451.8 [2327.5 to 5119.4] | 7801.4 [5724.2 to 10632.4] | 6547.7 [4589.9 to 9340.5] | 7265.8 [5028.1 to 10499.3] | 3334.0 [2310.7 to 4810.5]

22. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0 to Day 3) post-vaccination period
Population: The Booster Total Vaccinated cohort included all subjects vaccinated during the Booster stage, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 248 | 122 | 79 | 41 | 124
Participants
  Any Pain | 206 | 90 | 61 | 31 | 87
  Grade 3 Pain | 55 | 18 | 15 | 6 | 22
  Any Redness | 142 | 68 | 44 | 19 | 55
  Grade 3 Redness | 5 | 1 | 0 | 0 | 5
  Any Swelling | 114 | 48 | 38 | 20 | 51
  Grade 3 Swelling | 3 | 3 | 2 | 0 | 4

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite, fever [defined as axillary temperature equal to or above 38.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 248 | 122 | 79 | 41 | 124
Participants
  Any Drowsiness | 159 | 71 | 46 | 24 | 58
  Grade 3 Drowsiness | 1 | 2 | 1 | 0 | 4
  Related Drowsiness | 159 | 71 | 46 | 24 | 58
  Any Irritability | 198 | 89 | 58 | 29 | 79
  Grade 3 Irritability | 14 | 3 | 4 | 2 | 8
  Related Irritability | 198 | 89 | 58 | 29 | 79
  Any Loss of appetite | 130 | 54 | 32 | 19 | 57
  Grade 3 Loss of appetite | 6 | 3 | 0 | 0 | 2
  Related Loss of appetite | 130 | 54 | 32 | 19 | 57
  Any Fever | 133 | 56 | 43 | 20 | 55
  Grade 3 Fever | 21 | 6 | 7 | 4 | 11
  Related Fever | 133 | 56 | 43 | 20 | 55

24. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The Booster Total Vaccinated cohort included all subjects vaccinated during the Booster stage.
Measure: Count of Participants; unit: Participants
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 249 | 123 | 79 | 41 | 125
Participants | 7 | 4 | 0 | 2 | 8

25. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to one month Post-Booster vaccination
Population: The Booster Total Vaccinated cohort included all subjects vaccinated during the Booster stage.
Measure: Count of Participants; unit: Participants
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
Number analyzed (Participants) | 249 | 123 | 79 | 41 | 125
Participants | 8 | 0 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day (Days 0-3) post-booster vaccination period. Unsolicited AEs: within the 31-day (Days 0-30) post-booster vaccination period. SAEs: up to one month post-booster dose (Visit 2).
Arm/Group | ACAC GROUP | ACHibPS GROUP | HibACPS GROUP | HibHibPS GROUP | CC GROUP
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/123 | 0/79 | 0/41 | 0/125
Serious Adverse Events (participants affected / at risk) | 8/249 | 0/123 | 1/79 | 1/41 | 1/125
Other Adverse Events (participants affected / at risk) | 234/249 | 115/123 | 75/79 | 38/41 | 113/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACAC GROUP (N=249) | ACHibPS GROUP (N=123) | HibACPS GROUP (N=79) | HibHibPS GROUP (N=41) | CC GROUP (N=125)
Febrile convulsion (Nervous system disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACAC GROUP (N=249) | ACHibPS GROUP (N=123) | HibACPS GROUP (N=79) | HibHibPS GROUP (N=41) | CC GROUP (N=125)
Decreased appetite (Metabolism and nutrition disorders) | 130 (130) | 54 (54) | 32 (32) | 19 (19) | 57 (57)
Erythema (Skin and subcutaneous tissue disorders) | 142 (142) | 68 (68) | 44 (44) | 19 (19) | 55 (55)
Irritability (Psychiatric disorders) | 198 (198) | 89 (89) | 58 (58) | 29 (29) | 79 (79)
Pain (General disorders) | 206 (206) | 90 (90) | 61 (61) | 31 (31) | 87 (87)
Pyrexia (General disorders) | 135 (135) | 57 (57) | 43 (44) | 20 (20) | 56 (57)
Somnolence (Nervous system disorders) | 159 (159) | 71 (71) | 46 (46) | 24 (24) | 58 (58)
Swelling (General disorders) | 114 (114) | 48 (48) | 38 (38) | 20 (20) | 51 (51)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 7 (7) | 2 (2) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.